CLINICAL TRIAL: NCT01417507
Title: Natural History of Postoperative Cognitive Function, Quality of Life, and Seizure Control in Patients With Supratentorial Low-Risk Grade II Glioma
Brief Title: Natural History of Brain Function, Quality of Life, and Seizure Control in Patients With Brain Tumor Who Have Undergone Surgery
Status: Completed | Type: Observational
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: RTOG 0925; NCI-2011-02982 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000708271; U10CA037422 (NIH)
Record Dates: First submitted 2011-08-13; First posted 2011-08-16 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Adult Diffuse Astrocytoma; Adult Mixed Glioma; Adult Oligodendroglioma; Cognitive/Functional Effects; Neurotoxicity; Psychosocial Effects of Cancer and Its Treatment; Seizure
MeSH Terms: conditions — Astrocytoma; Glioma; Oligodendroglioma; Neurotoxicity Syndromes; Seizures | interventions — Mental Status and Dementia Tests; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue will be submitted to the RTOG Biospecimen Resource for the purpose of central review of pathology (mandatory fo eligibility), tissue banking, and translational research (highly recommended). For central review, H&E slide and tumor block must be submitted. For tissue banking and translational research, remaining tissue from the central review will be used and plasma, whole blood and urine will be collected.

GROUPS / COHORTS (1):
- Supportive care (neurocognitive assessment and MRI): Patients undergo neurocognitive assessment using the CogState Test battery (the DET, the IDN, the OCLT, and the GMLT) at baseline* and at 12, 24, 36, 42, 48, 54, and 60 months. Patients also complete the EORTC QOL-30, the BCM20, and the EQ-5D questionnaires at baseline*, at 12, 24, 36, 48, and 60 months afterwards, and before undergoing any further treatment. Patients are instructed to complete a seizure and medication diary during study.
  Patients undergo MRI scans at baseline*, at 12, 24, 36, 48, and 60 months, and at the time of radiological, clinical, or neurological failure.
  Interventions: Procedure: cognitive assessment; Procedure: magnetic resonance imaging; Other: laboratory biomarker analysis; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: cognitive assessment — Undergo neurocognitive assessment
Procedure: magnetic resonance imaging — Undergo MRI
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This trial studies the natural history of brain function, quality of life, and seizure control in patients with brain tumor who have undergone surgery. Learning about brain function, quality of life, and seizure control in patients with brain tumor who have undergone surgery may help doctors learn more about the disease and find better methods of treatment and on-going care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if there is difference in the average changes of neurocognitive function (NCF) scores from baseline to the time of radiologic tumor progression or up to 5 years (whichever occurs first), between radiologically progressed and non-progressed patients.

SECONDARY OBJECTIVES:

I. To determine if there is difference in the time to neurocognitive decline, as defined by the Reliable Change Index - Within subjects Standard Deviation (RCI-WSD), between radiologically progressed and non-progressed patients.

II. To evaluate NCF during the postoperative observational period of progression-free survival (PFS) and after radiological progression for a total time on study of 5 years.

III. To determine if the changes in cognitive functioning are an early warning biomarker for radiological progression.

IV. To explore the effect of salvage therapy on cognitive outcomes in patients who progress during the study period for up to 5 years.

V. To evaluate quality-of-life (QOL) as measured by the European Organization for Research and Treatment of Cancer (EORTC) QOL-30 and QOL brain module (BCN20) and health utilities as measured by the European Quality of Life-5 Dimensions (EQ-5D), for a total time on study of 5 years.

VI. To evaluate seizure control for a total time on study of 5 years. VII. To evaluate molecular correlates of QOL, NCF, seizure control, and PFS. VIII. To characterize aberrant molecular pathways in low-grade gliomas (LGGs) and test the hypothesis that activation of signaling pathways will predict worse PFS and overall survival (OS).

IX. To explore the relationship between change in cognitive function and symptomatic progression (defined as worsening seizures or new or progressive neurologic deficits) or clinical progression (defined as initiation of treatment interventions such as radiotherapy, chemotherapy, or additional surgery).

OUTLINE:

Patients undergo neurocognitive assessment using the CogState Test battery (the Detection Test (DET), the Identification Test (IDN), the One Card Learning Test (OCLT), and the Groton Maze Learning Test (GMLT)) at baseline* and at 12, 24, 36, 42, 48, 54, and 60 months. Patients also complete the EORTC Quality of Life Questionnaire-Core 30 (QOL-30), the Brain Cancer Module-20 (BCM20), and the European Quality of Life-5 Dimensions (EQ-5D) questionnaires at baseline*, at 12, 24, 36, 48, and 60 months afterwards, and before undergoing any further treatment. Patients are instructed to complete a seizure and medication diary during study.

Patients undergo MRI scans at baseline*, at 12, 24, 36, 48, and 60 months, and at the time of radiological, clinical, or neurological failure.

NOTE: * 12 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Central pathology confirmed diagnosis of supratentorial grade II oligodendroglioma, astrocytoma, or mixed oligoastrocytoma prior to step 2 registration
* No multifocal disease, based upon the following minimum diagnostic work-up:

  * History/physical examination, including neurologic examination, within 84 days prior to step 2 registration
  * Brain MRI with and without contrast within 84 days prior to Step 2 registration (Note: MRI 70 days after surgery is preferred and highly encouraged)
* The patient must be within one of the following categories:

  * Maximal safe resection with minimal residual disease defined as follows:

    * Removal of T2/fluid-attenuated inversion recovery (FLAIR) abnormalities thought to be primarily tumor, with a residual ≤ 2 cm maximal tumor diameter/T2 FLAIR abnormality on MRI to be done within 84 days post-operatively
    * If there is > 2 cm post-operative residual T2/FLAIR abnormality and the neurosurgeon believes this represents edema and not primarily tumor, the neurosurgeon is encouraged to repeat imaging within the allowed study period (up to 84 days post-operatively) to confirm resolution of edema

      * MRI at the time of enrollment must document a ≤ 2 cm residual maximal tumor diameter/T2 FLAIR abnormality
    * Patients who required a second surgery to obtain a maximal safe resection will be eligible if the second surgery is performed within 84 days of the initial diagnostic procedure
  * Age < 40 (any extent of resection)
  * Age < 50 and preoperative tumor diameter < 4 cm (any extent of resection)
* Karnofsky performance status ≥ 80%
* No prior invasive malignancy (except non-melanomatous skin cancer) unless disease-free for a minimum of 3 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Must be able to undergo MRI of the brain with gadolinium
* No plans for adjuvant radiotherapy or chemotherapy after surgery
* No more than 84 days (12 weeks) since prior surgery
* No brain tumor recurrence
* No prior brain tumor surgery, radiation therapy and/or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Central pathology-confirmed diagnosis of supratentorial grade II oligodendroglioma, astrocytome or mixed oligoastrocytoma prior to Step 2 registration.
  The patient must be within one of the following categories:
  Maximal safe resection with minimal residual disease defined as follows:
  * Removal of T2/FLAIR abnormalities thought to be primarily tumor, with a residual ≤ 2 cm maximal tumor diameter/T2 FLAIR abnormality on MRI to be done within 84 days postoperatively.
  * Patients who require a second surgery to obtain a maximal safe resection will be eligible if the second surgery is performed within 84 days of the inital diagnostic procedure.
  OR Age <40 (any extent of resection) OR Age <50, preoperative tumor diameter <4 cm (any extent of resection)
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
NCF as measured by each of the 4 neurocognitive tests (DET, IDN, OCLT, GMLT) | Up to 5 years
  Each of the battery's tests will be evaluated using the 2-sample t-test with a 2-sided significance level of 0.05 to determine if there is a clinically meaningful difference in the average change of NCF score from baseline to the time of radiologic tumor progression or up to 5 years (whichever occurs first) between radiologically progressed and non-progressed patients. In order to adjust for multiple comparisons and maintain the overall type I error of 0.05, Hochberg's procedure will be applied.

SECONDARY OUTCOMES:
Time to neurocognitive decline in patients who progress and who do not progress radiologically, as defined by the RCI-WSD | Up to 5 years
  The cumulative incidence approach will be used to estimate the median time to neurocognitive impairment to account for the competing risk of death and to determine if there is a clinically meaningful difference in the time to neurocognitive decline, as defined by the RCI-WSD (reliable change index-within-subjects standard deviation), between radiologically progressed and non-progressed patients.
PFS | The interval from registration to progression or death, whichever occurs first, assessed up to 5 years
  Estimated using the Kaplan-Meier method, and difference between the activation of different signaling pathways will be tested using the log rank test. Multivariate analyses with the Cox proportional hazards model for PFS will be performed to assess the activation of the signaling pathway effect adjusting for patient-specific risk factors. The covariates to be evaluated for the multivariate models are: activation of signaling pathway status, age, tumor size, and other prognostic factors.
Radiological progression | Up to 5 years
  To determine if the NCF decline is an earlier warning biomarker to radiologic progression, we will use NCF change as a time-dependent covariate in a Cox proportional hazards (PH) regression model with radiological progression as the endpoint. The Cox model estimates the ratio of hazard rate of radiographic failure with and without neurocognitive decline. Anticonvulsant use, tumor size, tumor histology, and further treatment received if recurrence is discovered, which may also have impact on the radiological progression, will also be considered in this Cox PH regression analysis.
Effect of salvage therapy on cognitive outcomes in patients who progress | Up to 5 years
QOL as measured by the EORTC QOL-30, EORTC QOL-BCN20, and EQ-5D | Up to 5 years
  The general linear mixed-effects model will be used to evaluate the changes of QOL and health utilities over time.
Frequency of seizures, evaluated using patient seizure diary | Up to 5 years
  Marginal models will be used to evaluate the change of frequencies of seizures over time for up to 5 years. Anticonvulsant use, tumor size, tumor histology, further treatment received if recurrence is discovered, and other prognostic factors will also be included in the covariates sets. The available molecular marker information will also be included as a covariate to evaluate the molecular correlates of seizure frequency.
Molecular correlates of QOL, NCF, seizure control, and PFS | Up to 5 years
OS | Up to 5 years
  Estimated using the Kaplan-Meier method, and difference between the activation of different signaling pathways will be tested using the log rank test. Multivariate analyses with the Cox proportional hazards model for OS will be performed to assess the activation of the signaling pathway effect adjusting for patient-specific risk factors. The covariates to be evaluated for the multivariate models are: activation of signaling pathway status, age, tumor size, and other prognostic factors.
Symptomatic or clinical progression | Up to 5 years
  Symptomatic and clinical progression will be explored for the correlation with cognitive changes in addition to radiological progression.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Choucair, Principal Investigator — Radiation Therapy Oncology Group
Locations (41):
- United States (39):
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Arizona Oncology-Deer Valley Center, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Florida Hospital, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - Hawaii Medical Center East, Honolulu, Hawaii
  - Leeward Radiation Oncology Center, ‘Ewa Beach, Hawaii
  - Evanston CCOP-NorthShore University HealthSystem, Evanston, Illinois
  - Covenant Medical Center, Waterloo, Iowa
  - Norton Health Care Pavilion - Downtown, Louisville, Kentucky
  - Norton Suburban Hospital, Louisville, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Barnes West County Hospital, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - The Nebraska Medical Center, Omaha, Nebraska
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Radiation Therapy Oncology Group, Philadelphia, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (2):
  - London Regional Cancer Program, London, Ontario
  - McGill University Department of Oncology, Montreal, Quebec